CLINICAL TRIAL: NCT03112668
Title: Couple-Focused ACT Intervention for Couples Coping With Cancer: A Pilot Study
Brief Title: Acceptance and Commitment Therapy in Improving Well-Being in Patients With Stage III-IV Cancer and Their Partners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sharon Manne, PhD, Professor of Medicine, Rutgers Cancer Institute of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro20170000115; NCI-2017-00445 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro20170000115; 131604 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2017-03-28; First posted 2017-04-13 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Malignant Female Reproductive System Neoplasm; Malignant Hepatobiliary Neoplasm; Partner; Stage III Breast Cancer; Stage III Cervical Cancer; Stage III Colorectal Cancer; Stage III Lung Cancer; Stage III Prostate Cancer; Stage III Skin Melanoma; Stage III Uterine Corpus Cancer; Stage IIIA Breast Cancer; Stage IIIA Cervical Cancer; Stage IIIA Colorectal Cancer; Stage IIIA Lung Carcinoma; Stage IIIA Skin Melanoma; Stage IIIA Uterine Corpus Cancer; Stage IIIB Breast Cancer; Stage IIIB Cervical Cancer; Stage IIIB Colorectal Cancer; Stage IIIB Lung Carcinoma; Stage IIIB Skin Melanoma; Stage IIIB Uterine Corpus Cancer; Stage IIIC Breast Cancer; Stage IIIC Colorectal Cancer; Stage IIIC Skin Melanoma; Stage IIIC Uterine Corpus Cancer; Stage IV Breast Cancer; Stage IV Cervical Cancer; Stage IV Colorectal Cancer; Stage IV Lung Cancer; Stage IV Prostate Cancer; Stage IV Skin Melanoma; Stage IV Uterine Corpus Cancer; Stage IVA Cervical Cancer; Stage IVA Colorectal Cancer; Stage IVA Uterine Corpus Cancer; Stage IVB Cervical Cancer; Stage IVB Colorectal Cancer; Stage IVB Uterine Corpus Cancer
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Melanoma | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (ACT) (Experimental): Patients and their partners attend 6 weekly ACT sessions over 60-75 minutes. Couples learn skills of acceptance, avoidance, awareness, values and committed action, mindfulness and values in relationships, and handling persistent worries and concerns. Patients and their partners also do homework assignment after each session.
  Interventions: Behavioral: Cognitive Behavior Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Survey Administration

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy — Undergo ACT
  Other Names: CBT; cognitive therapy; CT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies how well acceptance and commitment therapy works in improving well-being in patients with stage III-IV cancer and their partners. Learning how to accept negative thoughts and feelings and how to live in the present without worrying about the future or past may improve coping skills in patients with stage III-IV cancer and their partners.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the feasibility and acceptability of couples' acceptance and commitment therapy (ACT) (C-ACT).

II. To collect pilot data on the impact of C-ACT on patients' and partners' anxiety, depression, and quality of life.

OUTLINE:

Patients and their partners attend 6 weekly ACT sessions over 60-75 minutes. Couples learn skills of acceptance, avoidance, awareness, values and committed action, mindfulness and values in relationships, and handling persistent worries and concerns. Patients and their partners also do homework assignment after each session.

After completion of the study, patients and their partners are followed up at 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stage 3 or 4 breast, cervical, colorectal, endometrial, hepatobiliary, lung, melanoma, gynecological, prostate cancer in the past six months
* Married or cohabiting with a significant other of either gender for more than one year
* At the time of recruitment, a life expectancy of greater than 6 months and/or a Karnofsky performance status of 80 or above or an Eastern Cooperative Oncology Group (ECOG) score of 0 or 1
* English speaking
* No significant hearing impairment that would prevent participation in sessions
* Live within a 1 hour commuting distance from Rutgers Cancer Institute of New Jersey

Exclusion Criteria:

* Partner cannot have cancer diagnosis (other than non-melanoma skin cancer) and be currently receiving treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-01-25 (Actual)

PRIMARY OUTCOMES:
Change in acceptance as measured by the COPE acceptance subscale | Baseline to 1-week post intervention
  Pre-post changes will be examined using t-tests in the primary outcomes as well as the mechanisms of change (e.g., flexibility, avoidance self-disclosure). Because this is primarily a pilot and feasibility study and not an efficacy test, these data will be used primarily to examine whether an impact on distress and well-being was made but statistical significance will not be the primary aim.
Change in avoidance as measured by the Acceptance and Action Questionnaire-II | Baseline to 1-week post intervention
  Pre-post changes will be examined using t-tests in the primary outcomes as well as the mechanisms of change (e.g., flexibility, avoidance self-disclosure). Because this is primarily a pilot and feasibility study and not an efficacy test, these data will be used primarily to examine whether an impact on distress and well-being was made but statistical significance will not be the primary aim.
Change in value based living as measured by the Valued Living questionnaire | Baseline to 1-week post intervention
  Pre-post changes will be examined using t-tests in the primary outcomes as well as the mechanisms of change (e.g., flexibility, avoidance self-disclosure). Because this is primarily a pilot and feasibility study and not an efficacy test, these data will be used primarily to examine whether an impact on distress and well-being was made but statistical significance will not be the primary aim.
Feasibility defined as acceptance | Up to 1-week post intervention
  This trial will be considered feasible if the acceptance rate among eligible patients is equal to or greater than 30%
Feasibility defined as session drop out | Up to 1-week post intervention
  This trial will be considered feasible if drop out from sessions (at any point over the 6 sessions) is less than 20% (thus, 6/30)
Feasibility defined as survey follow ups | Up to 1-week post intervention
  This trial will be considered feasible if 3) completion of study surveys at the follow up is 80%, and patients are not lost to progressive disease.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Manne, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States